CLINICAL TRIAL: NCT05387200
Title: A Multi Center, Randomized, Open-label, Parallel, Phase IV Clinical Trial to Evaluate Efficacy and Safety of MASI BONE S (Alendronate Sodium Trihydrate) in Postmenopausal Women With Osteoporosis
Brief Title: Phase IV Clinical Trial to Evaluate Efficacy and Safety of MASI BONE S (Alendronate Sodium Trihydrate) in Postmenopausal Women With Osteoporosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0486
Record Dates: First submitted 2022-05-18; First posted 2022-05-24 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Masibone S (Experimental): Masibone S (alendronate sodium trihydrate 70mg, oral solution) 1 bottle weekly and cholecalciferol 1000U/calcium 100mg 1T daily for 48 weeks
  Interventions: Drug: Masibone S
- Fosamax (Active Comparator): Fosamax (aledronate sodium 70mg, oral tablet) 1T weekly and cholecalciferol 1000U/calcium 100mg 1T daily for 48 weeks
  Interventions: Drug: Fosamax

INTERVENTIONS:
Drug: Masibone S — The investigators will evaluate the change of bone mineral density at lumbar spine measured by DEXA after 48 weeks of alendronate sodium trihydrate 70mg (oral solution) 1 bottle weekly and cholecalciferol 1000U/calcium 100mg 1T daily use.
  Arms: Masibone S
Drug: Fosamax — The investigators will evaluate the change of bone mineral density at lumbar spine measured by DEXA after 48 weeks of alendronate sodium 70mg (oral tablet) 1T weekly and cholecalciferol 1000U/calcium 100mg 1T daily use.
  Arms: Fosamax

SUMMARY:
This study aims to prove non-inferiority of the efficacy of Masibone S (alendronate sodium trihydrate 70mg, oral solution) on the treatment of postmenopausal osteoporosis compared to the efficacy of Fosamax (alendronate sodium 70mg, oral tablet). The effect of Masibone S and Fosamax on bone mineral density in postmenopausal women with osteoporosis will be compared and analyzed. This study included a total 170 patients (85 per subgroup) for multi-center, randomized, open-label, parallel clinical trial. The drugs will be maintained for a total of 48 weeks. The primary endpoint is the difference of bone mineral density change at lumbar spine measured by DEXA between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. postmenopausal women ≥50 years old
2. osteoporosis - BMD T-score ≤-2.5 at lumbar spine, femoral neck, or total hip within previous 24 weeks

   - BMD T-score -1.0~-2.5 at lumbar spine, femoral neck, or total hip within previous 24 weeks and history of osteoporotic fractures - BMD T-score -1.0~-2.5 at lumbar spine, femoral neck, or total hip within previous 24 weeks and FRAX MOF >20% or HF >3%
3. Those who voluntarily agree in written form to participate in the clinical trial after hearing the explanation of this clinical trial and those who do not have any of exclusion criteria

Exclusion Criteria:

1. Patient with history of drugs that affect bone mineral density - bisphosphonate, denosumab, teriparatide, romosozumab within one year - calcitonin or analogues, calcimimetics within previous 12 weeks - strontium or fluoride for treating osteoporosis at any time in the past
2. Patients with history of osteonecrosis of jaw, osteonecrosis of external ear canal, or atypical femoral fracture
3. Patients with history of invasive dental procedure (tooth extraction, implant, oral surgery etc) within previous 24 weeks or patients who plan for invasive dental procedure during the clinical trial period
4. Patients with risk of aspiration (esophageal disorders such as esophageal stricture, achalasia or patients who can not sit or stand for more than 30 minutes)
5. Patients with severe renal dysfunction (eGFR by MDRD <30 ml/min/1.73m2 or on dialysis) or liver dysfunction (AST or ALT ≥x3 upper limit of normal reference range)
6. Patients who are under treatment or plan for treatment due to solid tumor or hematologic malignancy
7. Patients with secondary osteoporosis (persistent systemic steroid use, uncontrolled hyperthyroidism, primary hyperparathyroidism)
8. Hypocalcemia (albumin-corrected calcium <2.1mmol/L) or vitamin D deficiency (25OHD <10ng/mL) during screening
9. Patients with known allergic reaction, hypersensitivity, or intolerance to bisphosphonate and other components of intervention drugs during screening (including latex allergy and hereditary fructose intolerance)
10. Patients who the examiner considers not eligible for clinical trials

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Enrollment: 170 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Change of bone mineral density at lumbar spine | 48 weeks
  DEXA is used to evaluate the change of bone mineral density at lumbar spine after 48 weeks of drug intervention compared to those at baseline

SECONDARY OUTCOMES:
Change of serum levels of bone turnover markers | 24 and 48 weeks
  Serum levels bone turnover markers (CTX and P1NP) is measured at baseline and after 24 and 48 weeks of drug intervention and the change of serum levels of CTX and P1NP is evaluated.
Adherence to drug | 24 and 48 weeks
  The proportion of patients who compliantly uses drugs after 24 and 48 weeks of intervention will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yumie Rhee, Principal Investigator — Department of Internal Medicine, Endocrine Research Institute, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baek S, Ahn SH, Hong N, Seo DH, Hong S, Rhee Y. Efficacy and safety of weekly liquid alendronate in Korean postmenopausal women with osteoporosis: a 12-month, multi-center, randomized trial. Arch Osteoporos. 2024 Nov 26;19(1):119. doi: 10.1007/s11657-024-01480-6. PMID 39589664